CLINICAL TRIAL: NCT01691157
Title: The Effectiveness of Exercise in the Physiotherapy Management of Subacromial Impingement Syndrome
Brief Title: Exercise in the Physiotherapy Management of Shoulder Impingement
Acronym: EaSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ulster (Other)
Collaborators: Belfast Health and Social Care Trust (Other); Northern Health and Social Care Trust (Other Government); Mayo Clinic (Other); Keele University (Other)
Responsible Party: Principal Investigator, Dr Joseph G McVeigh, Lecturer in Physiotherapy and PhD supervisor, University of Ulster
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11/NI/0026 version 3.1
Record Dates: First submitted 2012-08-08; First posted 2012-09-24 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Subacromial Impingement Syndrome
Keywords: Subacromial impingement syndrome; Rotator cuff; Exercise; Physiotherapy
MeSH Terms: conditions — Shoulder Impingement Syndrome; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual physiotherapy without exercise (Active Comparator): Will receive 6 sessions of modified usual physiotherapy care that can consist of any physiotherapeutic modalities normally provided except exercise. this may consist of postural advice, taping, electrotherapy, acupuncture, manual joint mobilizations of the shoulder, cervical or thoracic spine.
  Interventions: Other: Usual physiotherapy without exercise
- Exercise (Experimental): Will receive an evidence based exercise protocol but no other physiotherapeutic modalities
  Interventions: Other: Evidence based exercise protocol

INTERVENTIONS:
Other: Evidence based exercise protocol — An evidence based graduated exercise rehabilitation protocol will be provided and supervised by a physiotherapist. patients will receive 6 sessions of supervised physiotherapy
  Arms: Exercise
Other: Usual physiotherapy without exercise — Will receive modified usual physiotherapy care that can consist of any physiotherapeutic modalities normally provided except exercise. this may consist of postural advice, taping, electrotherapy, acupuncture, manual joint mobilizations of the shoulder, cervical or thoracic spine.
  Other Names: Usual care
  Arms: Usual physiotherapy without exercise

SUMMARY:
The purpose of this trial is to investigate the effectiveness of an evidence based exercise program for shoulder impingement. Approximately 1% of adults consult their General Practitioner (GP) with shoulder pain each year, making it the third most common reason for musculoskeletal GP consultations in the UK. A further 50% of these patients are diagnosed with subacromial impingement syndrome (SAIS) (shoulder impingement syndrome) and commonly referred for physiotherapy treatment. This trial aims to compare the effectiveness of an evidence based exercise protocol with usual physiotherapy care.

DETAILED DESCRIPTION:
Physiotherapy management of shoulder impingement frequently involves exercise, however there is little evidence underpinning exercise prescription and outcomes are poor. Few trials have investigated which muscles should be targeted and how they should be strengthened with respect to the mode, frequency, duration, intensity and progression. This is a randomized controlled trial(RCT) investigating the effectiveness of an evidence based exercise program for shoulder impingement. This research may have an impact on how physiotherapists provide exercise programs to patients with shoulder impingement.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be aged 18 years and older.
* Shoulder pain of at least 3/10 in severity that has been diagnosed by a consultant rheumatologist, orthopaedic surgeon or general practitioner within the past 12 months.
* Positive Hawkins-Kennedy test.
* Positive on testing either supraspinatus (empty can test) or infraspinatus (resisted external rotation in neutral).

Exclusion Criteria:

* Acute traumatic conditions.
* Evidence of rotator cuff tear (positive drop arm test) or any other shoulder joint pathology (e.g. adhesive capsulitis, labral tears).
* A history of fractures of the upper arm, shoulder or clavicle within the past two years.
* A history of dislocation of the shoulder within the previous two years.
* Postoperative conditions involving the upper arm, shoulder or clavicle.
* Inflammatory or systemic diseases.
* Current signs and symptoms of acute nerve root pain arising from the cervical or upper thoracic spine.
* Previous physiotherapy for the same condition involving an exercise regime.
* Previous corticosteroid injection of the affected shoulder within the past 6 months.
* Unwilling participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
change from baseline in average pain scores at rest and at night using 100mm visual analogue scale (VAS). | Outcomes measured at 0, 6 and 12 weeks
  Primary outcome measure: Average pain scores at rest and at night for the week prior to measurement will be recorded using a 100mm visual analogue scale (VAS). The change in pain scores at 6 and 12 weeks from baseline will be measured.

SECONDARY OUTCOMES:
Western Ontario Rotator Cuff Index (WORC | 0, 6 and 12 weeks
  Secondary outcome measures will focus on function, disability and quality of life, consisting of a combination of generic, region specific and disease-specific health questionnaires. The change in scores from baseline will be measured.
The American Shoulder and Elbow Surgeons function score. | 0. 6 and 12 weeks
  Limb specific outcome measure
SF-36 Health Survey • SF-36 Health Survey | 0, 6 and 12 weeks
  Generic measure of health status
Isometric strength and range of movement of shoulder flexion, abduction, external rotation and internal rotation using a hand held dynamometer. | 0, 6 and 12 weeks
  objective measures of strength and ROM

CONTACTS AND LOCATIONS:
Overall Officials: Joseph G McVeigh, BSc Hons, Principal Investigator — University of Ulster
Locations (4):
- United Kingdom (4):
  - Musgrave Park Hospital, Belfast, N.Ireland
  - The Waveney Hospital, Ballymena, N.I
  - Robinson Memorial Hospital, Ballymoney, N.I
  - The Fort Centre, Physiotherapy Department, Coleraine, N.I